CLINICAL TRIAL: NCT07258147
Title: Clinical Study on the Efficacy and Safety of Radiotherapy Combined With Immunotherapy and Chemotherapy for Pre-treated Patients With Small Cell Lung Cancer and Liver Metastases
Brief Title: Safety and Efficacy of Radiotherapy Combined With Immunochemotherapy in Pre-treated SCLC Patients With Liver Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Division of Thoracic Tumor Multimodality Treatment, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLC-LM-001
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (SCLC)
Keywords: SCLC; Radiotherapy; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy; Drug Therapy; Etoposide; 130-nm albumin-bound paclitaxel; Irinotecan; PM 01183; Radiation; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation therapy combined with immunotherapy and chemotherapy group (Experimental): Liver-directed radiotherapy (low-dose radiation(3Gy*5d) or low-dose radiation(3Gy*5d) +stereotactic body radiation therapy (10Gy*3d) ) followed by immunotherapy combined with chemotherapy (Etoposide, Nab-paclitaxel, Irinotecan, or Lurbinectedin) administered systemically every 3 weeks. Immunotherapy is continued as maintenance therapy until disease progression or for up to 24 months.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy (Etoposide, Nab-paclitaxel, Irinotecan, or Lurbinectedin); Radiation: low-dose radiation; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Immunotherapy — Combined With Chemotherapy( (Etoposide, Nab-paclitaxel, Irinotecan, or Lurbinectedin) ). Liver-directed radiotherapy (low-dose radiation(3Gy*5d) or low-dose radiation(3Gy*5d) +stereotactic body radiation therapy (10Gy*3d) ) followed by Immunotherapy
Drug: Chemotherapy (Etoposide, Nab-paclitaxel, Irinotecan, or Lurbinectedin) — Combined With immunotherapy.
Radiation: low-dose radiation — Liver-directed radiotherapy (low-dose radiation(3Gy*5d) followed by Immunotherapy
Radiation: Stereotactic Body Radiation Therapy (SBRT) — low-dose radiation(3Gy*5d) +stereotactic body radiation therapy (10Gy*3d) )

SUMMARY:
This is clinical trial evaluating the safety and efficacy of radiotherapy combined with immunotherapy and chemotherapy in patients with extensive-stage small-cell lung cancer (ES-SCLC) and liver metastases.

DETAILED DESCRIPTION:
All eligible patients will receive liver-directed radiotherapy, followed by PD-1/PD-L1 inhibitors plus chemotherapy. The systemic therapy is initiated concurrently with radiotherapy. PD-1/PD-L1 inhibitors and chemotherapeutic agents (such as Etoposide, Nab-paclitaxel, Irinotecan, or Lurbinectedin) are administered intravenously every 3 weeks according to their approved product information. The treatment regimen consists of an initial concurrent phase of radiotherapy, immunotherapy, and chemotherapy, followed by a maintenance phase with PD-1/PD-L1 inhibitors alone until disease progression or for up to 24 months.Main Objective and Endpoint:

The primary objective is to evaluate the objective response rate (ORR) and safety of the combination therapy. The primary endpoint is the ORR, defined as the proportion of subjects achieving a complete response (CR) or partial response (PR) based on RECIST v1.1 criteria, as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, with an ECOG Performance Status of 0-2.
2. Histologically confirmed stage IV non-small cell lung cancer (NSCLC) or extensive-stage small cell lung cancer, with radiologically confirmed liver metastases (at least one measurable lesion with the longest diameter ≥ 1 cm).
3. Prior failure (due to progression or intolerance) to platinum-based doublet chemotherapy and PD-1/PD-L1 inhibitor therapy.
4. Adequate liver function reserve (Child-Pugh class A or B, ALT/AST ≤ 5 × ULN, total bilirubin ≤ 1.5 × ULN).
5. Life expectancy of at least 3 months.
6. Normal function of major organs and no severe dysfunction of the hematopoietic, cardiac, pulmonary, hepatic, renal, or bone marrow systems, or immunodeficiency diseases.
7. Within one week prior to enrollment, bone marrow and organ function meet the following criteria:Hemoglobin ≥ 80 g/L, neutrophil count ≥ 1.5 × 10⁹/L, and platelet count ≥ 70 × 10⁹/L. Renal function: Serum creatinine ≤ 1.5 × ULN, and endogenous creatinine clearance rate ≥ 55 ml/min.Liver function: Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN (if liver metastases are present, total bilirubin ≤ 3 × ULN and transaminases ≤ 5 × ULN are acceptable).
8. Voluntarily participates and provides written informed consent.
9. Good compliance and willingness to adhere to the study visit schedule and other protocol requirements.
10. Willingness to provide blood and tissue samples for biomarker testing.
11. Judged by the radiation oncologist to have no contraindications to liver radiotherapy. Patients who agree to receive immunotherapy, chemotherapy, and radiotherapy.
12. For patients of childbearing potential: agreement to use effective contraception during the study period and for at least 6 months after the last study treatment; negative serum or urine pregnancy test within 7 days prior to study entry; and not breastfeeding. Male patients with partners of childbearing potential must agree to use effective contraception during the study and for 6 months after the last dose.

Exclusion Criteria:

1. Presence of any active autoimmune disease or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism [may be included if controlled with hormone replacement therapy]); prior liver radiotherapy or liver transplantation; history of liver cirrhosis (Fibroscan ≥ F3), portal hypertension, or hepatic encephalopathy.
2. Congenital or acquired immunodeficiency, such as Human Immunodeficiency Virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive HCV antibody and HCV RNA above the lower limit of detection of the assay), or co-infection with both hepatitis B and C.
3. Uncontrolled or significant cardiac disease, including: (a) NYHA Class II or higher heart failure; (b) Unstable angina; (c) Myocardial infarction within the past 1 year; (d) Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
4. Severe infection or serious comorbidities within 4 weeks prior to the first dose of study treatment.
5. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
6. History of other primary malignancies within the past 5 years.
7. Known allergy to any of the trial drugs or their excipients.
8. Pregnant or lactating women, or subjects of childbearing potential unwilling to use effective contraception during the study period.
9. Patients with Child-Pugh class B or C liver insufficiency.
10. Any other contraindication as determined by the investigator to preclude participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of enrollment until the first documented date of disease progression or death from any cause (whichever occurs first), assessed up to 24 months.
  The proportion of participants who achieve a best overall response of Complete Response (CR) or Partial Response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as assessed by the investigator.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment until first progression or death, assessed up to approximately 3 years.
  The time from the date of enrollment until the first documented date of disease progression as per RECIST v1.1, or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | From enrollment until the first documented date of disease progression, assessed up to 24 months.
  The proportion of participants who achieve a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST v1.1.
Incidence of Adverse Events (AEs) | From the first dose of study treatment until 30 days after the last dose (up to approximately 25 months).
  The number and percentage of participants with any adverse event, serious adverse event, and immune-related adverse event. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, Principal Investigator — Principal Investigator
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen Z, Wu L, Wang Q, Yu Y, Liu X, Ma R, Li T, Li Y, Song X, Li L, Zhao W, Wang Q, Xu X, Lu S. Brief Report: Ivonescimab Combined With Etoposide Plus Carboplatin as First-Line Treatment for Extensive-Stage SCLC: Results of a Phase 1b Clinical Trial. J Thorac Oncol. 2025 Feb;20(2):233-239. doi: 10.1016/j.jtho.2024.10.013. Epub 2024 Oct 28. PMID 39490738
- [Result] Wang H, Yao Z, Kang K, Zhou L, Xiu W, Sun J, Xie C, Yu M, Li Y, Zhang Y, Zheng Y, Lin G, Pan X, Wu Y, Luo R, Wang L, Tang M, Liao S, Zhu J, Zhou X, Zhang X, Xu Y, Liu Y, Peng F, Wang J, Xiang L, Yin L, Deng L, Huang M, Gong Y, Zou B, Wang H, Wu L, Yuan Z, Bi N, Fan M, Xu Y, Tong R, Yi L, Gan L, Xue J, Mo X, Chen C, Na F, Lu Y. Preclinical study and phase II trial of adapting low-dose radiotherapy to immunotherapy in small cell lung cancer. Med. 2024 Oct 11;5(10):1237-1254.e9. doi: 10.1016/j.medj.2024.06.002. Epub 2024 Jul 3. PMID 38964333